CLINICAL TRIAL: NCT03110536
Title: Sindromul de Burnout la asistenții Medicali de Triaj Din unitățile de Primire urgențe
Brief Title: The Burnout Syndrome in Emergency Department Triage Nurses
Acronym: BurN_ED
Status: Completed | Type: Observational
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Collaborators: County Clinical Emergency Hospital Cluj-Napoca (Other)
Responsible Party: Principal Investigator, Eugenia-Maria Muresan, Principal Investigator, Iuliu Hatieganu University of Medicine and Pharmacy
Other Study IDs: 9253/11.04.2017
Record Dates: First submitted 2017-04-07; First posted 2017-04-12 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Burnout, Professional; Nurse's Role
Keywords: Burnout syndrome; Triage; Nurse; Emergency Department; Romania
MeSH Terms: conditions — Burnout, Professional; Burnout, Psychological; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 2h assessment: The assessment of the burnout syndrome will be carried out at the beginning of the triage shift and after 2 hours.
  Interventions: Diagnostic Test: Copenhagen Burnout Inventory; Other: Triage scoring efficacy
- 4h assessment: The assessment of the burnout syndrome will be carried out at the beginning of the triage shift and after 4 hours.
  Interventions: Diagnostic Test: Copenhagen Burnout Inventory; Other: Triage scoring efficacy
- 6h assessment: The assessment of the burnout syndrome will be carried out at the beginning of the triage shift and after 6 hours.
  Interventions: Diagnostic Test: Copenhagen Burnout Inventory; Other: Triage scoring efficacy

INTERVENTIONS:
Diagnostic Test: Copenhagen Burnout Inventory — A questionnaire based on Copenhagen Burnout Inventory will be completed by each participant to the study, at the beginning of the triage shift and after 2, 4 or 6 hours.
  The questionnaire also contains clinical cases that require triage coding.
Other: Triage scoring efficacy — The triage scores of the first 5 and the last 5 cases assessed by the investigated nurse will be compared with the triage codes of an expert evaluator (nurse involved in designing The National triage Protocol).

SUMMARY:
Assessment of burnout syndrome of triage nurses from Emergency Departments from Cluj-Napoca, Romania.

DETAILED DESCRIPTION:
This study is aiming at assessing the burnout syndrome amongst triage nurses working in the Emergency Departments in Cluj-Napoca. The study design is observational, prospective and multicentric.

At this moment, there are 43 nurses covering triage shifts in the Emergency Clincial County Hospital Cluj and 18 more within Emergency Clinical Hospital for Children Cluj-Napoca. On average, these ED roughly attend 90.000 patients yearly.

Questionnaires are based on Copenhagen Burnout Inventory, with additional clinical cases that require triage coding according to The Romanian National Triage Protocol of 2016. Each triage nurse will complete the questionnaire when beginning the triage shift and after a period of 2, 4 or 6 hours.

ELIGIBILITY:
Inclusion Criteria:

* ED nurse within Emergency Clinical County Hospital Cluj and Emergency Clinic Hospital for Children Cluj-Napoca.

Exclusion Criteria:

* triage experience of at least 1 year

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Emergency Department nurses from Emergency Clinical County Hospital Cluj and Emergency Clinic Hospital for Children Cluj-Napoca.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Assessment of burnout syndrome in triage ED nurses | 2 to 6 hours
  Copenhagen Burnout Inventory

SECONDARY OUTCOMES:
Efficacy of triage ED nurses | 2 to 6 hours
  The triage scores of the first 5 and the last 5 cases assessed by the investigated nurse will be compared with the diagnostic codes of the physicians who treated those patients.

CONTACTS AND LOCATIONS:
Locations (2):
- Romania (2):
  - Emergency County Hospital for Children, Cluj-Napoca, Cluj
  - Emergency Clinical County Hospital Cluj-Napoca - Emergency Department, Cluj-Napoca, Cluj

IPD SHARING:
Plan to Share IPD: No